CLINICAL TRIAL: NCT02605096
Title: A Single Centre Randomised, Non-blinded, Prospective Pilot to Test the Feasibility Associated With the Use of MRI as the Initial Imaging Modality in the Investigation of Patients Presenting With Suspected Scaphoid Fracture
Brief Title: Pilot Study to Test the Feasibility of the Use of MRI in Suspected Scaphoid Fractures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment strategy not working. This information was really useful to design a randomised controlled trial.
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RJ115/N294
Record Dates: First submitted 2015-11-05; First posted 2015-11-16 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Scaphoid Fracture
Keywords: suspected scaphoid fracture
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MRI group (Experimental): This arm assess the use of MRI as the first line examination of suspected scaphoid fracture (replacing conventional plain x-ray).
  Patients with negative findings will receive a splint and contact card to a specialist wrist clinic if the pain persists for ten to fourteen days after initial presentation.
  Patients with positive findings will receive a plaster cast and undergo a CT scan (to evaluate displacement) and will be referred to the fracture clinic. Furthermore, if the CT scan confirms a displaced fracture, that might require surgery, the patient should be seen by a Hand Specialist at fracture clinic.
  All patients enrolled in the pilot should undergo a 4-view plain x-ray 3 months after the initial ED/UCC presentation.
  Interventions: Procedure: MRI
- X-ray group (Active Comparator): This arm is the current standard of care pathway for the diagnosis of patients with suspected scaphoid fracture. This includes an initial clinical assessment on arrival to the Emergency Department of Urgent Care Centre followed by a plain x-ray (using a 4-view scaphoid protocol).
  Patients with negative/positive findings for scaphoid fracture in the initial X-ray will be immobilised with a splint/plaster cast.
  All patients will be referred to an initial fracture clinic and a proportion of patients are likely to require additional imaging scans (usually CT but also MRI) and follow-up appointments in the fracture clinic. All patients enrolled in the pilot should undergo a 4-view plain x-ray 3 months after the initial ED/UCC presentation.
  Interventions: Procedure: X-ray

INTERVENTIONS:
Procedure: MRI — Magnetic Resonance Imaging Scan
  Arms: MRI group
Procedure: X-ray — X-ray exam (conventional radiography)
  Arms: X-ray group

SUMMARY:
This pilot study aims to test the feasibility and work flows associated with using MRI as the initial imaging modality in the investigation of patients presenting with suspected scaphoid fracture.

This pilot will be used to inform the design of a study that will aim to evaluate whether the proposed intervention is likely to generate cost-savings whilst improving or maintaining overall patient quality of life and satisfaction.

DETAILED DESCRIPTION:
The present pilot study is designed to assess the feasibility of using MRI as the initial imaging modality in the investigation of patients presenting with suspected scaphoid fracture at the Emergency department or Urgent Care Centre. This study will inform the design of a study that will aim to evaluate whether the proposed intervention is likely to generate cost-savings whilst improving or maintaining overall patient quality of life and satisfaction.

Patients with a suspected scaphoid fracture will be randomised to receive standard of care using 4-view plain x-ray (control group) as the first imaging modality or MRI examination as the first imaging modality.

ELIGIBILITY:
Inclusion Criteria:

* Patients considered to be suitable for the proposed pathway include every patient aged 16 years old or above, presenting at A&E/UCC between 8:00am and 4:00pm (Monday to Friday), with at least one of the following:
* Isolated pain / tenderness over the Anatomical Snuff Box (ASB) or scaphoid tubercle or pain in the scaphoid region during axial loading of the 1st metacarpal.
* History of recent fall (< 14 days) on out-stretched hand (FOOSH), wrist injury or poor history associated with examination findings suggestive of scaphoid fracture.

Exclusion Criteria:

* Patients presenting outside GSTT's catchment area not willing to be followed-up at GSTT;
* Patients without suspected scaphoid fracture following an initial A&E/UCC clinical triage;
* Patients with scaphoid fracture not admitted through A&E at St Thomas' Hospital or Urgent Care Centre at Guy's Hospital;
* Patients presenting at ED/UCC on weekdays (Monday to Friday) before 8:00am or after 4:00pm
* Patients presenting at ED/UCC on weekends or Bank Holidays;
* Patients who lack capacity to give consent or participate in the study;
* Patients that are already taking part in a clinical trial of an investigational medicinal products (CTIMPs);
* Patient is unable or unsuitable to MRI

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-04-01 (Actual)

PRIMARY OUTCOMES:
Time elapsed (measured in hours and minutes) from A&E presentation to study recruitment. | 1 month
  Please note that the submitted study is a pilot to test feasibility of main study. Due to the recruitment of patients from A&E, informed consent will need to be obtained for the study without negatively impacting clinical care (E.g Delay to treatment of patient with scaphoid fracture).
Recruitment rate | 1 month
  Number of patients recruited divided by total number of patients eligible and approached
The proportion of mandatory fields of the Case Report Form completed including eligibility criteria, medical examination and history, patient demographics, randomisation and documents checklist. | 1 month
  This will test the study's data collection procedures.
Time elapsed (measured in hours and minutes) from A&E presentation to the initial MRI or x-ray investigation. | 1 month
Time elapsed (measured in hours and minutes) from A&E presentation to treatment (either plaster cast or removable splint). | 1 month
Time elapsed (measured in hours and minutes) from A&E presentation to A&E discharge. | 1 month

SECONDARY OUTCOMES:
Study attrition rate | 4 months
  % patients lost to follow-up
The proportion of patient who completed the EQ-5D-5L questionnaire. | 4 months
  Data collected will be used to inform the main study and will determine if any change in processes is required, prior to commencing main study.
The proportion of patient who completed the patient resource use diary. | 4 months
  Data collected will be used to inform the main study and will determine if any change in processes is required, prior to commencing main study.
The proportion of patient who completed the patient experience questionnaire. | 4 months
  Data collected will be used to inform the main study and will determine if any change in processes is required, prior to commencing main study.

CONTACTS AND LOCATIONS:
Overall Officials: sanjay vijayanathan, MRCP FRCR, Principal Investigator — Guy's and St Thomas Hospital NHS Foundation